CLINICAL TRIAL: NCT02570334
Title: A Cross Sectional Evaluation of the Development in Children Age 4 to 7 Infected or Exposed to HIV From the ANRS 12140 Cohort (Pediacam)
Acronym: PediacamDEV
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: ANRS, Emerging Infectious Diseases (Other Government)
Collaborators: Centre Pasteur du Cameroun (Other); Hopital Universitaire Robert-Debre (Other); Institut de Recherche pour le Developpement (Other Government); Centre Mère et Enfant de la Fondation Chantal Biya (Other); Hospital General De Douala (Other); Centre Hospitalier D'essos (Other); Inserm U1018, Equipe 4 VIH & IST (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: ANRS 12322 PediacamDEV
Record Dates: First submitted 2015-10-06; First posted 2015-10-07 (Estimated); Last update posted 2016-07-12 (Estimated); Status verified 2016-07

CONDITIONS: HIV; HIV-uninfected Children; Children Exposed to HIV
Keywords: early ART; neurocognitive evaluation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- HIV-infected children diagnosed before 7 months of life (Experimental): HIV-infected children diagnosed before 7 months of life
  Interventions: Other: HIV-infected children initiated antiretroviral treatment within the first 7 months of life
- HIV-exposed uninfected children (Experimental): HIV-uninfected children born to HIV-infected mothers
  Interventions: Other: HIV-infected children initiated antiretroviral treatment within the first 7 months of life
- HIV-unexposed uninfected children (Experimental): Children born to HIV-uninfected mothers
  Interventions: Other: HIV-infected children initiated antiretroviral treatment within the first 7 months of life

INTERVENTIONS:
Other: HIV-infected children initiated antiretroviral treatment within the first 7 months of life — All arms will recieve a thourough clinical evaluation : Global motor development (Touwen test), global cognitive development (K-ABC II test), visual (Log Mar Char) and hearing (full ear nose and throat examination) impediments as well as a questionnaire concerning socioeconomic situation, medical history of the child and mother, and HIV treatment and follow up information.

SUMMARY:
This study aims to perform a comprehensive neuro-cognitive evaluation of the 4-7 year old children from the Pediacam cohort (ANRS 12140 /12225, NCT02043418). It is expected thereby to provide complementary information to the trials CHER and PREDICT on the long term development of (1) HIV-infected children according to age at ARV initiation and (2) HIV exposed but not infected children, all compared with the control group of children uninfected, unexposed to HIV.

DETAILED DESCRIPTION:
Cognitive, motor and sensorial impairments associated to HIV infection have been and remain important concerns in children. The advent of ARV has reduced the frequency and the extent of HIV-related encephalopathys, but literature suggests that more limited impairments remain (CHER and PREDICT trials). These neuro-cognitive disorders might constitute an important public health problem in sub-Saharan Africa where a high percentage of children born to HIV+ women live. Nevertheless,the knowledge on their long-term consequences on children development in this context remains limited. Data on the burden of cognitive, motor and sensorial impairment in resource-limited settings as well as on the interaction with other factors that could also impair children development are scarse.

The Pediacam cohort gives the opportunity to better understand the development of children born to HIV-infected mothers - infected by HIV or not - followed up from birth and living in sub-Saharan Africa.

ELIGIBILITY:
Inclusion Criteria:

* Children included in the Pediacam cohort and age 4 to 7
* Parent or guardian written informed consent obtained

Exclusion Criteria:

-

Ages: 4 Years to 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 400 (Estimated)
Dates: Start 2015-12; Primary Completion 2016-10 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Global motor development (Touwen test), global cognitive development (K-ABC II test), visual (Log Mar Char) and hearing (full ear nose and throat examination) impediments | 4-7 years of age
  Frequency of cognitive, motor and sensorial impairments in 4-7 year old children born to HIV+ mothers who received early treatment in the first 7 months of life

SECONDARY OUTCOMES:
Compared frequency of motor, cognitive and sensorial impairments between infected and uninfected children | 4-7 years of age
  long term effect of HIV and/or PMTCT exposure on children exposed but not infected with HIV. Results of cognitive, motor and sensorial (hearing and visual) evaluations will be compared among cohorts.
Effect of early ARV (<3 months) versus differed ARV (between 3 and 7 months) on neurocognitive impairments | 4-7 years of age
  long term effect of early ARV (<3 months) versus differed ARV (between 3 and 7 months) on cognitive, motor and sensorial impairments in HIV+ children
Prognostic factors and consequences of HIV-associated neuro-cognitive impairments | 4-7 years of age
  prognostic factors and describe consequences of HIV-associated neuro-cognitive impairments on children social life

CONTACTS AND LOCATIONS:
Locations (3):
- Cameroon (3):
  - Hôpital de Laquintinie, Douala
  - Centre Hospitalier d'Essos, Yaoundé
  - Hôpital de la Fondation Mère-enfant Chantal Biya, Yaoundé